CLINICAL TRIAL: NCT01010646
Title: Multicentre, Randomised, Open-label Study Comparing the Tolerability and Viral Reduction of the Combination of IFN Alpha-2b XL + Ribavirin Versus Peg IFN Alpha-2b + Ribavirin in Patients With Chronic Hepatitis C, Genotype 1 or 4.
Brief Title: Study Comparing the Tolerability and Viral Reduction of the Combination of IFN a-2b XL + Ribavirin Versus Peg IFN a-2b + Ribavirin in Patients With Chronic Hepatitis C, Genotype 1 or 4
Acronym: COAT IFN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Flamel Technologies (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-015121-37; ANRS HC 23 COAT-IFN
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Hepatitis C
Keywords: hepatitis C; viral kinetics; antiviral response; Genotype 1 or 4
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GP1N IFN alfa-2bXL 27 MUI + Ribavirin (Experimental): IFN alfa-2bXL 27 MUI, powder and solvent for solution injection
  Interventions: Drug: IFN alfa-2b XL 27 MUI + Ribavirin
- GP2N IFN alfa-2b XL 36 MUI + Ribavirin (Experimental): IFN alfa-2b XL 36 MUI, powder and solvent for solution injection
  Interventions: Drug: IFN alfa-2b XL 36 MUI + Ribavirin
- GP3N IFN peg alfa-2b 1.5 µg/kg + Ribavirin (Active Comparator): IFN peg alfa-2b 1.5 µg/kg,administered once a week for 12 weeks by subcutaneous injections
  Interventions: Drug: IFN peg alfa-2b 1.5 µg/kg + Ribavirin

INTERVENTIONS:
Drug: IFN alfa-2b XL 27 MUI + Ribavirin — IFN alfa-2b XL 27 MUI administered once a week for 12 weeks by subcutaneous injections, in combination with weight dosed ribavirin daily administered orally in two divided doses
  Arms: GP1N IFN alfa-2bXL 27 MUI + Ribavirin
Drug: IFN alfa-2b XL 36 MUI + Ribavirin — IFN alfa-2b XL 36 MUI administered once a week for 12 weeks by subcutaneous injections in combination with weight dosed ribavirin daily administered orally in two divided doses
  Arms: GP2N IFN alfa-2b XL 36 MUI + Ribavirin
Drug: IFN peg alfa-2b 1.5 µg/kg + Ribavirin — IFN peg alfa-2b 1.5 µg/kg administered once a week for 12 weeks by subcutaneous injections in combination with weight dosed ribavirin daily administered orally in two divided doses
  Arms: GP3N IFN peg alfa-2b 1.5 µg/kg + Ribavirin

SUMMARY:
Three-parallel-arm, open-label, international (France and Romania) study, comparing three treatments

The purpose of this study is to confirm if IFN alfa-2b XL has a better antiviral activity and tolerability as compared with current marketed reference, while combined with ribavirin, in a 3-month therapy setting.

DETAILED DESCRIPTION:
Interferon alfa-2b XL (IFN alfa-2b XL) is a novel sustained release interferon α-2b drug product that is being developed by FLAMEL TECHNOLOGIES using its Medusa® technology, aiming at reducing the toxicity and enhancing the biological response. In the present study, patients will be randomly assigned to either IFN alfa-2b XL 27 MUI, IFN alfa-2b XL 36 MUI, or IFN peg alfa-2b 1.5 µg/kg, all administered once a week for 12 weeks by subcutaneous injections, in combination with weight dosed ribavirin daily administered orally in two divided doses. Doses will be adapted according to the dose modification guidelines for combination therapy labelled in the ribavirin prescribing information.

ELIGIBILITY:
Inclusion Criteria:

* Patient having voluntarily signed the Informed Consent Form prior to any study specific procedure being performed
* Male or female HCV genotype 1 or 4 infected patients (positive serum HCV RNA), aged between 18 and 65 years inclusive, with a body mass within the range over or equal of 45Kg and below or equal to 100 Kg
* Patient being either naïve to therapy, either non-responder to previous standard Peg-interferon α + ribavirin therapy,
* With no absolute contra-indication to interferon α or ribavirin
* Female patients must be non-lactating and of non-childbearing potential, or have a negative pregnancy test results to enter the study
* No evidence of acute or advanced liver disease, uncontrolled diabetes, cardiovascular, immunological, or thyroid disease, and no recently diagnosed malignancy
* Vital signs within normal ranges, or if outside the normal ranges, not deemed clinically significant in the opinion of the Investigator. An ECG with no clinically significant abnormalities

Exclusion Criteria:

* History of solid organ transplantation
* Severe systemic infection, uncontrolled diabetes, cancers, associated liver disease
* General anesthesia or recent blood transfusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-09 (Actual); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Viral load decrease at Week 4 and Week 12 of treatment with IFN alfa-2b XL 27 MIU, IFN alfa-2b XL 36 MIU and the marketed reference product (PEG IFN alfa-2b 1.5μg/kg) in combination with ribavirin | Week 4 and Week 12

SECONDARY OUTCOMES:
Percentage of patients with early virologic response (EVR) (reduction of at least 2 log viral load) at the end of week 12 | Week 4 and Week 12
Percentage of patients with complete early virologic response (EVR) (viral load <15 IU) at the end of the week 12 | Week 4 and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Christian TREPO, MD, Principal Investigator — Hôpital de la Croix Rousse, Service d'Hépato-Gastro-Entérologie, 69004 Lyon - FRANCE
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- See also: French National Agency for Research on AIDS and Viral Hepatitis website — http://www.anrs.fr